CLINICAL TRIAL: NCT01505400
Title: Integrated Molecular Profiling in Advanced Cancers Trial
Acronym: IMPACT
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: IMPACT-001
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Non-small Cell Lung Cancer; Colorectal Cancer; Genitourinary Cancer; Pancreatobiliary Gastrointestinal Cancer; Upper Aerodigestive Tract Cancer; Gynecological Cancers; Melanoma Cancers; Rare Cancers; Unknown Primary Cancers
Keywords: Molecular profiling; Advanced cancer; Breast cancer; Non-small cell lung cancer; Colorectal cancer; Genitourinary cancer; Pancreatobiliary gastrointestinal cancer; Upper aerodigestive tract cancer; Gynecological cancers; Phase I; Phase I Clinical Trial Candidates; melanoma cancer; rare cancer; unknown primary cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Urogenital Neoplasms; Neoplasms, Unknown Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archival tumor tissue
  1 tube of whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced cancer: Advanced breast, non-small cell lung, colorectal, genitourinary, pancreatobiliary gastrointestinal, upper aerodigestive tract, gynecological, melanoma, unknown primary, and rare carcinomas; as well as patients who are phase I trial candidates

SUMMARY:
Substantial progress has been made in the treatment of cancer through the use of targeted therapies, but what works for one patient might not work for another patient. Certain drugs are now being developed that target specific molecules in the body that are believed to be part of the disease.

Biomarkers are specific characteristics of the cancer that may help provide prognostic information (i.e. how well patients will be regardless of the treatments given) or help predict sensitivity or resistance to a specific treatment.

The study will collect archival tumor samples (previously collected biopsy or surgical tumor samples) to provide biomarker data about a patient's cancer, in order to help their physicians to identify which clinical trials of molecularly targeted therapies may be most appropriate for the patient in the future.

DETAILED DESCRIPTION:
The increasing appreciation and identification of specific somatic mutations and other genetic aberrations that drive cancers leave us on the threshold of a new era of "personalized cancer medicine", in which specific biomarkers will be used to direct targeted agents only to those patients deemed most likely to respond. The potential medical, scientific and economic benefits of such a personalized approach to cancer therapy are immense and self-evident. Yet despite some important advances, only a limited number of approved targeted agents have had their approvals predicated on specific biomarkers of sensitivity or resistance.

The premises behind personalized cancer medicine include: i) genetic aberrations exist in human malignancies; ii) a subset of these aberrations, often present across multiple cancer types, have functional relevance as "hallmarks" or "drivers" for oncogenesis and tumor progression; iii) such genetic aberrations are potentially "druggable" targets; and iv) there are tolerable medicinal compounds that can effectively modulate such targets. A key requirement of this new, personalized approach to anti-cancer therapy is that specific patients must be matched to a particular drug or combination of drugs. Molecular profiling of tumors to identify somatic mutations and/or other genetic aberrations are examples of enrichment strategies to assist in matching patients to drugs or treatments that have gained increasing interest in the oncology community.

The present protocol seeks to provide molecular profiling data to the treating physician for patients with advanced breast, non-small cell lung, colorectal, genitourinary, pancreatobiliary gastrointestinal, upper aerodigestive tract, gynecological, melanoma, unknown primary, and rare carcinomas, as well as patients who are phase I trial candidates, in order to help identify which standard regimens or clinical trials of molecularly targeted therapies may be most appropriate for the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological confirmation of advanced breast, non-small cell lung, colorectal, genitourinary, pancreatobiliary gastrointestinal, upper aerodigestive tract, gynecological, melanoma, unknown primary, and rare carcinomas who are candidates for systemic therapy, as well as patients who are phase I trial candidates.
* Patient must be ≥ 18 years old.
* Patient's ECOG performance status equal to 0 or 1.
* All patients must have signed and dated an informed consent form.
* All patients must have sufficient archived tumor tissue for molecular profiling.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced cancers (breast, non-small cell lung, colorectal, genitourinary, pancreatobiliary gastrointestinal, upper aerodigestive tract, gynecological, melanoma, unknown primary, and rare carcinomas) and phase 1 clinical trial candidates
Sampling Method: Probability Sample
Enrollment: 3026 (Actual)
Dates: Start 2012-02; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Molecular profiling data to be made available in patient's electronic medical records. | 1 month
  Genotyping assays including: AKT1, HRAS, AKT2, JAK2, AKT3, KIT, BRAF, KRAS, CDK, MEK1, CTNNB1, MET, EGFR, NOTCH1, ERBB2, NRAS, FGFR1, PDGFRA, FGFR2, PIK3CA, FGFR3, RET, FGFR4, SMO, STK11

SECONDARY OUTCOMES:
Utilization rates of molecular profiling information | 1 year
  Including utilization of information for standard regimens or clinical trials of molecularly targeted therapies.
Clinical trial accrual rates among patients with available molecular profiling data | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bedard, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Ma LX, Espin-Garcia O, Bedard PL, Stockley T, Prince R, Mete O, Krzyzanowska MK. Clinical Application of Next-Generation Sequencing in Advanced Thyroid Cancers. Thyroid. 2022 Jun;32(6):657-666. doi: 10.1089/thy.2021.0542. Epub 2022 May 16. PMID 35262412
- [Derived] Stockley TL, Oza AM, Berman HK, Leighl NB, Knox JJ, Shepherd FA, Chen EX, Krzyzanowska MK, Dhani N, Joshua AM, Tsao MS, Serra S, Clarke B, Roehrl MH, Zhang T, Sukhai MA, Califaretti N, Trinkaus M, Shaw P, van der Kwast T, Wang L, Virtanen C, Kim RH, Razak AR, Hansen AR, Yu C, Pugh TJ, Kamel-Reid S, Siu LL, Bedard PL. Molecular profiling of advanced solid tumors and patient outcomes with genotype-matched clinical trials: the Princess Margaret IMPACT/COMPACT trial. Genome Med. 2016 Oct 25;8(1):109. doi: 10.1186/s13073-016-0364-2. PMID 27782854